CLINICAL TRIAL: NCT00173901
Title: Adverse Drug Reactions of Different Brands of Ceftazidime Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 900104
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2001-01

CONDITIONS: Infection
Keywords: ceftazidime; safety; infection
MeSH Terms: conditions — Infections | interventions — Ceftazidime

INTERVENTIONS:
Drug: ceftazidime

SUMMARY:
The purpose of this study is to understand whether generic ceftazidime causes different adverse drug reaction incidence from the brand drug.

DETAILED DESCRIPTION:
Ceftazidime is a third generation cephalosporins that should be reserved for severe bacterial infections. Substitution of the brand ceftazidime with a generic ceftazidime raised some concerns.

The purpose of this study is to understand whether generic ceftazidime causes different adverse drug reaction incidence from the brand drug.

ELIGIBILITY:
Inclusion Criteria:

* patients in surgical intensive care unit who require ceftazidime treatment

Exclusion Criteria:

* less than 1 year old

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 536
Dates: Start 2001-03; Study Completion 2002-04

PRIMARY OUTCOMES:
The adverse drug reactions of ceftazidime

SECONDARY OUTCOMES:
The effectiveness of ceftazidime

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Chwen Chang, MD PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan